CLINICAL TRIAL: NCT00643214
Title: A Study to Determine if Tetrix Cream Impedes the Resolution of Experimentally Induced Allergic Contact Dermatitis
Brief Title: Evaluation of Tetrix Cream in the Healing of Injured Skin in Subjects With Contact Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coria Laboratories, Ltd. (Industry)
Responsible Party: D. Innes Cargill, PhD, Coria Laboratories, Ltd.
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 806 805 09 003
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Tetrix Cream; Antigen reaction; effect on healing; To determine if application of Tetrix Cream to lesions of contact dermatitis interferes with their rate of healing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Twice daily topical application
  Interventions: Device: Tetrix
- 2 (Placebo Comparator): Twice daily topical application
  Interventions: Device: Tetrix

INTERVENTIONS:
Device: Tetrix — Twice daily topical application
  Arms: 1
Device: Tetrix — Twice daily topical application
  Arms: 2

SUMMARY:
To determine if Tetrix Cream,, when applied to the skin lesions on patients with contact dermatitis, slows or interferes with the healing of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects with sensitivity to nickel.

Exclusion Criteria:

* Under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Clearing of signs and symptoms of contact dermatitis | 10 days after induction of lesion and start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fowler, MD, Principal Investigator — Dermatology Specialists, LLC
Locations (1):
- Dermatology Specialists, LLC, Louisville, Kentucky, United States